CLINICAL TRIAL: NCT02664532
Title: Miller Straight Blade With Paraglossal Technique Compared to the Macintosh Blade in Respect to Visualization of Larynx and Ease of Intubation
Brief Title: Miller Straight Blade vs Macintosh Blade
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Main Hospital (Other)
Responsible Party: Principal Investigator, Dr.Deb Sanjay Nag, Associate Specialist, Tata Main Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: PR/JHTMH/09242A
Record Dates: First submitted 2016-01-10; First posted 2016-01-27 (Estimated); Results first posted 2016-03-11 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-02

CONDITIONS: Intubation; Difficult

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Miller group (Experimental): In Miller group, no 3 Miller blade was used for laryngoscopy by paraglossal technique. While intubating, the endotracheal tube (ETT) was directed underneath the laryngoscope blade without allowing it to go lateral to the blade. The curvature of the ETT automatically brings the tip towards the vocal cords as it was advanced. After successful endotracheal intubation, the ETT was attached to the circuit and anaesthesia continued as per plan.
  Interventions: Other: Miller group
- Macintosh group (Other): In Macintosh group, the curved blade was introduced to lift the base of the epiglottis to visualize larynx and then trachea intubated conventionally.After successful endotracheal intubation, the ETT was attached to the circuit and anaesthesia continued as per plan.
  Interventions: Other: Macintosh group

INTERVENTIONS:
Other: Miller group — Miller blade was used for laryngoscopy
  Arms: Miller group
Other: Macintosh group — Macintosh blade was used for laryngoscopy
  Arms: Macintosh group

SUMMARY:
The purpose of this prospective open labeled randomized study was to compare the "laryngoscopic glottis view" as well as "ease of intubation" between the two blades in routine intubations in non-difficult airways.

DETAILED DESCRIPTION:
One hundred and fifty patients with predicted non difficult airway were randomly assigned into two groups. After induction of anaesthesia laryngoscopy was performed with respective blades and trachea intubated. Parameters monitored were: glottis view obtained during laryngoscopy (Cormack Lehane grade), ease of intubation, intubation attempts, total duration of laryngoscopy in seconds and encountered complications.

ELIGIBILITY:
Inclusion Criteria:

* All ASA I & II grade patients undergoing elective surgery requiring general anesthesia with oral endotracheal intubation

Exclusion Criteria:

* Patients with anticipated difficult airway
* Cervical spine disorders
* Anesthesia requiring rapid sequence induction

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bhanu Pratap Swain, DNB, Principal Investigator — Tata Main Hospital, Jamshedpur,India

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Miller Group | Macintosh Group
Started | 75 | 75
Completed | 75 | 75
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: ASA grade I & II patients aged between 18 to 70 years of both genders undergoing elective surgery requiring general anesthesia with oral endotracheal intubation were included in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Miller Group | Macintosh Group | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 75 | 75 | 150
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (13.1) | 48.2 (14) | 47.6 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 47 | 93
  Male | 29 | 28 | 57
Region of Enrollment [Number; unit: participants] — All patients were from India (Jamshedpur)
  participants
    India | 75 | 75 | 150

OUTCOME MEASURES:

1. Primary Outcome: Ease of Intubation or Degree of Difficulty With Intubation
Description: Degree of difficulty with intubation Grade 1 Intubation easy Grade 2 Intubation requiring an increased anterior lifting force/optimal external laryngeal manipulation (OELM)/assistance to pull the right corner of the mouth upwards to augment space Grade 3 Intubation requiring more than one attempt or bougie guided intubation Grade 4 failure to intubate with the assigned laryngoscope
Time Frame: 60 seconds
Measure: Number; unit: participants
Arm/Group | Miller Group | Macintosh Group
Number analyzed (Participants) | 75 | 75
participants
  Grade 1 | 52 | 54
  Grade 2 | 23 | 16
  Grade 3 | 0 | 5
  Grade 4 | 0 | 0

2. Secondary Outcome: Cormack Lehane Grading
Description: Grade 1 Full view of glottis Grade 2 Only posterior commissure visible Grade 3 Only epiglottis visible Grade 4 No glottis structure visible
Time Frame: 60 seconds
Measure: Number; unit: participants
Arm/Group | Miller Group | Macintosh Group
Number analyzed (Participants) | 75 | 75
participants
  Grade 1 | 69 | 51
  Grade 2 | 6 | 18
  Grade 3 | 0 | 6
  Grade 4 | 0 | 0

3. Secondary Outcome: Number of Intubation Attempts
Description: An intubation attempt is defined as "intubation activities occurring during a single continuous laryngoscopy maneuver". Thus, even if several attempts were made to place an endotracheal tube during the course of a single laryngoscopy, this would be counted as a single intubation attempt.
Time Frame: 180 seconds
Measure: Number; unit: participants
Arm/Group | Miller Group | Macintosh Group
Number analyzed (Participants) | 75 | 75
participants
  Single Attempt | 75 | 74
  Second attempt | 0 | 1

4. Secondary Outcome: Total Laryngoscopy Duration in Seconds
Description: The duration of intubation was defined as the time taken from placement of the laryngoscope in the mouth to the time taken to remove the laryngoscope from the mouth following intubation.
Time Frame: 180 seconds
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Miller Group | Macintosh Group
Number analyzed (Participants) | 75 | 75
Seconds | 23 (7) | 20.5 (7.7)

ADVERSE EVENTS:
Time Frame: During the duration of admission in the hospital
Description: No adverse event was reported
Arm/Group | Miller Group | Macintosh Group
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/75
Other Adverse Events (participants affected / at risk) | 0/75 | 0/75

LIMITATIONS AND CAVEATS:
Blinding of laryngoscope to the laryngoscopist was not possible. The study was conducted in predicted non-difficult airways and cannot be extrapolated in difficult airway situations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes